CLINICAL TRIAL: NCT02179047
Title: Correlational Study on the Biomarkers Application to the Prediction and Diagnosis of Cardiovascular Diseases
Status: Completed | Type: Observational
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Yueh-Chung, Chen, chief of ICU, Taipei City Hospital
Other Study IDs: TCHIRB-1030509-E
Record Dates: First submitted 2014-05-27; First posted 2014-07-01 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2017-04

CONDITIONS: Stable Angina
Keywords: SYNTAX ,NGAL,Cystatin C,Galectin-3,Copeptin.MR-ProANP,sST2.
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ELISA kit for Human Galectin-3 Quantikine ELISA Kit (R&D system, Minneapolis, Mn)、Human ST2/IL-1 R4 Quantikine ELISA Kit(R&D system, Minneapolis, Mn)、Human Cystatin C Quantikine ELISA Kit(R&D system, Minneapolis, Mn)、 Human Lipocalin-2/NGAL Quantikine ELISA Kit(R&D system, Minneapolis, Mn)、Human midregional pro-atrial natriuretic peptide(MR-proANP) ELISA Kit(Cusabio, China, Cn)、Soluble ST2/IL-1R4 (HUMAN) Elisa Kit(AvisceraBioscience, Santa Clara,Ca)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- stable angina, biomarker: patients with stable angina who received coronary angiography.
  Interventions: Procedure: coronary angiography
- placebo: healthy subject
  Interventions: Procedure: coronary angiography

INTERVENTIONS:
Procedure: coronary angiography — percutaneous coronary intervention. coronary angiography.

SUMMARY:
Through the literature review , we pick out a series of forward-looking biological indicators as follows :

1. NGAL
2. Cystatin C:
3. Galectin-3:
4. Copeptin:
5. MR-Pro ANP:
6. sST2:

DETAILED DESCRIPTION:
1) NGAL (Neutrophil Gelatinase Associated Lipocalin): in the cardiovascular system , NGAL and endothelial cell apoptosis , atherosclerosis , and abdominal aortic aneurysm associated with thrombosis of a relationship. Heart and kidney complications in common a number of studies have demonstrated that NGAL in acute heart failure , cardiac catheterization / angiography management, and diagnostic usefulness of acute coronary artery disease and heart surgery , and how to make NGAL may pathological processes in the cardiovascular play a role. In the past studies have also demonstrated in sepsis (sepsis), cardiopulmonary around to support cardiac surgery, caused by acute renal developer injury and renal transplant patients and other studies confirm this early detection of serum creatinine more acute kidney injury . So we tried to make the results in this study .

(2) Cystatin C: Chronic kidney disease is a cardiovascular morbidity and mortality risk and a significant global health problem. Has been used to estimate renal function , serum creatinine, can be used instead . In several studies have shown to be more sensitive than that for predicting eGFRcreat serum creatinine or adverse events. This parameter also showed greater diagnostic sensitivity for the detection of mild renal damage . Cystatin C and metabolic syndrome and cardiovascular risk factors is also a correlation study confirmed (M. Magnusson et.al, 2013). Therefore , Cystatin C is emerging as a new biomarker for cardiovascular disease.

(3) Galectin-3: has proven to be a marker of myocardial fibrosis, Lars Gullestad , who in 2012 also found that Galectin-3 is mainly predictive of ischemic etiology . elderly patients with systolic heart failure death. And approved by the U.S. Food and Drug Administration to help in the prognosis of patients with heart failure in 2011 . Research has also pointed out that , Galectin-3 and there is a positive correlation between renal injury , and the correlation is not affected by whether the patients suffering from heart failure while affected.

(4) Copeptin: Copeptin was considered non -specific stress response of the marker , and may also have been proposed various non- cardiovascular monitoring and early warning and cardiovascular diseases ( coronary artery disease, heart failure and acute ) , etc., in a previous study , including patients with acute myocardial infarction was found with Copeptin related , and there Copeptin associated left ventricular ejection fraction (LVEF), and also the follow-up patients found to have a direct correlation with left ventricular volume, and is considered poor prognostic factor of death.

(5) MR-Pro ANP (midregional-Pro atrial natriuretic peptide): discovery and diagnosis of heart failure can be predicted in 1984, is a major discovery in the field of biological indicators of heart , but also a milestone, Elif Elmas et al found that when the 2011 MR-Pro ANP in patients suffering from cardiovascular disease as a diagnosis of myocardial fibrosis new biological indicators. Past research has also pointed out that can be used to predict lower respiratory tract infections and pneumonia, long and short-term mortality, Alzheimer's disease, and can diagnose sepsis and bacterial shock and prognosis prediction .

(6) sST2 (somatostatin2): Excessive sST2 may cause abnormal cardiac hypertrophy , fibrosis, and heart failure . Clinically, symptoms of heart failure with a high concentration of the patients diagnosed with sST2 severity determined correlations to predict increased risk of complications. Past research indicates measured values sST2 patients suffering from cardiovascular disease increased Jie phenomenon, and found that the measured values sST severity of cardiovascular disease 2 was positively correlated, has now been approved for use in patients with cardiovascular disease and new biomarkers predictive value of heart failure and death , but for the progress of heart failure severity change , changes in the measured value for sST2 correlation someone has not been confirmed.

ELIGIBILITY:
Inclusion Criteria:

* stable angina who eligible for coronary angiography after non-invasive stress test.

Exclusion Criteria:

* intolerance to procedure or contarst medium.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with stable angina who received coronary angiography.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: patients with stable angina who received coronary angiography and percutaneous coronary intervention.
- Placebo: healthy subjects
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 194 | 20
Completed | 187 | 20
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stable Angina: receive coronary angiogram
- Total: Total of all reporting groups
Arm/Group | Stable Angina | Placebo | Total
Number analyzed (Participants) | 187 | 20 | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 137 | 14 | 151
  >=65 years | 50 | 6 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (14) | 60 (12) | 61 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 6 | 56
  Male | 137 | 14 | 151
Region of Enrollment [Number; unit: participants]
  Taiwan | 187 | 20 | 207

OUTCOME MEASURES:

1. Primary Outcome: Biomarker Titer of Patients With Coronary Artery Disease
Description: The titer of 6 biomarkers(NGAL,Cystatin C,Galectin-3,Copeptin,MR-Pro ANP,sST2).
Time Frame: 6-12 months
Measure: Geometric Mean (95% Confidence Interval); unit: tilter
Units Other Than Participants: lesions
Groups:
- NGAL; Cystatin C; Galectin-3; Copeptin; MR-Pro ANP; sST2: biomarker
Arm/Group | NGAL | Cystatin C | Galectin-3 | Copeptin | MR-Pro ANP | sST2
Number analyzed (Participants) | 187 | 187 | 187 | 187 | 187 | 187
Number analyzed (lesions) | 187 | 187 | 187 | 187 | 187 | 187
tilter | 13 [2 to 36] | 5 [0 to 10] | 60 [1 to 120] | 0.5 [0.024 to 0.76] | 0.16 [0.008 to 0.26] | 184 [9 to 218]
Statistical Analysis 1: Comparison: NGAL vs Cystatin C vs Galectin-3 vs Copeptin vs MR-Pro ANP vs sST2; Test type: Superiority; p = 0.002, ANOVA; Hazard Ratio (HR) = 1.02

2. Primary Outcome: Biomarker of Healthy Subjects(Placebo)
Description: The relationship of 6 biomarkers(NGAL,Cystatin C,Galectin-3,Copeptin,MR-Pro ANP,sST2) of healthy subjects(placebo).
Time Frame: 6-12 months
Measure: Geometric Mean (95% Confidence Interval); unit: tilter
Units Other Than Participants: lesions
Arm/Group | NGAL | Cystatin C | Galectin-3 | Copeptin | MR-Pro ANP | sST2
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Number analyzed (lesions) | 20 | 20 | 20 | 20 | 20 | 20
tilter | 12 [1 to 34] | 4 [1 to 12] | 52 [2 to 82] | 0.1 [0.01 to 0.4] | 0.12 [0.09 to 0.83] | 121 [68 to 178]
Statistical Analysis 1: Comparison: NGAL vs Cystatin C vs Galectin-3 vs Copeptin vs MR-Pro ANP vs sST2; Test type: Superiority; p = 0.002, ANOVA; Hazard Ratio (HR) = 1.05, Standard Deviation 0.005

3. Primary Outcome: SYNTAX(SYNergy Between Percutaneous Coronary Intervention With TAXus) for Stable Angina Receveived Coronary Angiogram
Description: The relationship of 6 biomarkers(NGAL,Cystatin C,Galectin-3,Copeptin,MR-Pro ANP,sST2) with SYNTAX score.
  The SYNTAX Score is a unique tool to score complexity of coronary artery disease; there is no theoretical range existed for the SYNTAX score.
  Low risk:<22; intermediate risk: 22-33, high risk:>33
Time Frame: 6-12 months
Population: The SYNTAX Score is a unique tool to score complexity of coronary artery disease; there is no theoretical range existed for the SYNTAX score.
  SYNTAX Web site: http://www.syntaxscore.com/index.php Low risk:<22; intermediate risk: 22-33, high risk:>33
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: lesions
Groups:
- NGAL; Cystatin C; Galectin-3; Copeptin; MR-Pro ANP; sST2: patients with stable angina who received coronary angiography.
- Placebo(Healthy Subjects): patients without stable angina who received coronary angiography.
Arm/Group | NGAL | Cystatin C | Galectin-3 | Copeptin | MR-Pro ANP | sST2 | Placebo(Healthy Subjects)
Number analyzed (Participants) | 187 | 187 | 187 | 187 | 187 | 187 | 187
Number analyzed (lesions) | 187 | 187 | 187 | 187 | 187 | 187 | 187
scores on a scale | 22 (8) | 19 (4) | 32 (8) | 28 (13) | 33 (15) | 19 (3) | 6 (2)
Statistical Analysis 1: Comparison: NGAL vs Cystatin C vs Galectin-3 vs Copeptin vs MR-Pro ANP vs sST2; Test type: Superiority; p = 0.001, ANCOVA; Hazard Ratio (HR) = 1.39, Standard Deviation 0.005

ADVERSE EVENTS:
Groups:
- Intervention; Placebo: patients with worsen of angina symptoms after percutaneous coronary intervention.
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/187 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/187 | 0/20
Other Adverse Events (participants affected / at risk) | 0/187 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes